CLINICAL TRIAL: NCT03396250
Title: An Open Label Crossover Pharmacokinetic Trial of Naproxen Sodium and Diphenhydramine Hydrochloride Soft Capsules Versus Naproxen Sodium and Diphenhydramine Hydrochloride Tablets in Healthy Adult Subjects Under Fasted Conditions
Brief Title: A Pharmacokinetic Trial of Naproxen Sodium and Diphenhydramine Hydrochloride Soft Capsules Versus Naproxen Sodium and Diphenhydramine Hydrochloride Tablets in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17934
Record Dates: First submitted 2018-01-05; First posted 2018-01-10 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test product + Reference product (Experimental): Each treatment sequence consists of two treatment periods with each period consisting of 4 days starting with an overnight fast of at least 10 hours followed by a single dose of study drug administration the morning of Day 1, then a 72-hour PK (Pharmacokinetic) blood sampling period. The two drug administrations are separated by a 7 calendar days washout phase.
  Interventions: Drug: Naproxen sodium and diphenhydramine hydrochloride soft capsules; Drug: Naproxen sodium and diphenhydramine hydrochloride coated tablets (Aleve, PMBAY98-7111)
- Reference product + Test product (Experimental): Each treatment sequence consists of two treatment periods with each period consisting of 4 days starting with an overnight fast of at least 10 hours followed by a single dose of study drug administration the morning of Day 1, then a 72-hour PK blood sampling period. The two drug administrations are separated by a 7 calendar days washout phase.
  Interventions: Drug: Naproxen sodium and diphenhydramine hydrochloride soft capsules; Drug: Naproxen sodium and diphenhydramine hydrochloride coated tablets (Aleve, PMBAY98-7111)

INTERVENTIONS:
Drug: Naproxen sodium and diphenhydramine hydrochloride soft capsules — Single oral administration of Naproxen sodium 220 mg/DPH HCl 25mg (2 capsules)
Drug: Naproxen sodium and diphenhydramine hydrochloride coated tablets (Aleve, PMBAY98-7111) — Single administration of Naproxen sodium 220 mg/DPH HCl 25mg (2 tablets)

SUMMARY:
To evaluate the relative bioavailability of Naproxen Sodium 220 mg and diphenhydramine hydrochloride (DPH HCL) 25 mg soft capsules (Test) versus Naproxen Sodium 220 mg and diphenhydramine hydrochloride 25 mg tablets (Reference) after a single oral administration under fasted condition in healthy adults subjects.

To assess the safety and tolerability of the investigational products in terms of advent events (AEs) and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men or women
* Age 18 to 55 years inclusive;
* Body mass index 18.5 to 30.0 kg/m2 inclusive

Exclusion Criteria:

* History of hypersensitivity symptoms with the use of naproxen/naproxen sodium, diphenhydramine hydrochloride/citrate, acetylsalicylic acid, other Nonsteroidal anti-inflammatory drugs (NSAIDs) or similar pharmacological agents or components of the products;
* Females who are pregnant or lactating;
* Vegetarian or restricted diet (e.g., gluten-free);
* Any active disease, acute or chronic;
* Have taken naproxen/naproxen sodium, DPH HCl or diphenhydramine citrate, DPH HCl or diphenhydramine citrate-containing products, acetylsalicylic acid (ASA), ASA-containing products, acetaminophen, ibuprofen, any other NSAID (Over-the -counter [OTC] or prescription) or NSAID containing products, xanthines, antihistamines or caffeine-containing products (e.g. coffee, tea and chocolate) 7 days prior to dosing or during the Dosing Periods, other than trial treatment;
* Use of any over-the-counter or prescription medications, vitamins or herbal supplements (except acceptable forms of birth control) within 7 days prior to dosing or throughout the trial, unless in the opinion of the Investigator, the medication will not interfere with the trial procedures, data integrity, or compromise the safety of the subject;
* Positive test for Human immunodeficiency virus (HIV) antibodies and antigens;
* Positive test for hepatitis B surface antigen (HBsAg) test;
* Positive test for anti-hepatitis C virus (Anti-HCV) antibodies;
* In the judgment of the investigator, any need of other medication during the trial besides the test and reference study medication;
* Recently had (past 30 days) or plan to have surgery, an invasive procedure, tattoos or piercings during the trial or within 2 weeks after treatment;
* More than moderate alcohol consumption (>40 g of alcohol regularly per day);
* Positive alcohol or drug screen at Screening or on Day -1 of each dosing period.
* Any history or suspicion of barbiturate, amphetamine, benzodiazepine, cocaine, opiates, methamphetamine or cannabis abuse;
* Loss of blood in excess of 50 mL to 499 mL within 30 days or 500 ml within 56 days of the first dose of trial treatment (e.g., donation, plasmapheresis or injury);
* Excessive sports or sauna within 5 days before start of the treatment phase and unwilling to abstain during the trial;
* Have a platelet count <150,000/mm3 and in the judgment of the investigator, presents a significant bleeding risk;
* History of gastrointestinal bleeding or perforation, related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding);
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases (including glaucoma or benign prostatic hypertrophy) or malignancies or any other disease or condition which could influence the metabolism of the drug;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
AUC | Within 30 minutes prior to dosing (baseline) 10, 20, 30, 45, 60 minutes and 1 hour 20 minutes, 1 hour 40 minutes, 2, 2 hours 30 minutes, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose
  Area under the concentration vs. time curve from zero to infinity after single (first) dose
AUC(0-tlast) | Within 30 minutes prior to dosing (baseline) 10, 20, 30, 45, 60 minutes and 1 hour 20 minutes, 1 hour 40 minutes, 2, 2 hours 30 minutes, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose
  Area under plasma concentration vs. time curve from zero to last data point >LLOQ (lower limit of quantitation), calculated up by linear trapezoidal rule, down by logarithmic trapezoidal rule
Cmax | Within 30 minutes prior to dosing (baseline) 10, 20, 30, 45, 60 minutes and 1 hour 20 minutes, 1 hour 40 minutes, 2, 2 hours 30 minutes, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36, 48 and 72 hours post-dose
  Maximum observed drug concentration, directly observed from analytical data

SECONDARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | Up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- ICON Development Solutions, LLC, San Antonio, Texas, United States